CLINICAL TRIAL: NCT06645366
Title: Evaluation of Safety and Efficacy of the BTL-785F Device for Improvement in Skin Quality and Texture on Face and Neck
Brief Title: Device for Improving Skin Quality and Texture on the Face and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS1700
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-10

CONDITIONS: Wrinkle; Pigmentation; Skin Laxity; Skin Scarring
Keywords: skin; texture; wrinkles; skin quality
MeSH Terms: conditions — Cutis Laxa; Cicatrix | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with BTL-785F (Experimental): Three (3) treatment sessions will be applied to the subjects' face and neck using the BTL-785F system.
  Interventions: Device: Treatment with BTL-785F

INTERVENTIONS:
Device: Treatment with BTL-785F — Three (3) treatment sessions will be applied to the subjects' face and neck using the BTL-785F system equipped with the BTL-785-4-4 tip on BTL-785-4 applicator, lasting from 20 to 60 minutes depending on the size of the treated area. Each treatment will be spaced 2 - 6 weeks apart, after the complete healing of scabs.

SUMMARY:
The goal of this clinical trial is to investigate the effect of the BTL-785F device (with BTL-785-4-4 tip on BTL-785-4 applicator) on the improvement of skin quality and texture on the face and neck in healthy adult volunteers. The main question it aims to answer is:

Whether the BTL-785F device (with BTL-785-4-4 tip on BTL-785-4 applicator) is able to improve skin quality 3 months post-treatment, as assessed by two-dimensional and three-dimensional photographs.

Participants will complete three treatments, and two follow-up visits.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of the BTL-785F system equipped with the BTL-785-4-4 tip on BTL-785-4 applicator for the improvement of skin quality and texture on the face and neck. It is a prospective, multi-center, open label, one-arm study.

Subjects will be required to complete three (3) treatment visits and two (2) follow-up visits (at 1 month, 3 months post-treatment).

At baseline, inclusion and exclusion criteria will be verified upon obtaining informed consent from the patient. 2D and 3D photographs of the subjects will be taken.

The treatment administration phase consists of three (3) treatment visits, delivered 2 - 6 weeks apart, after the complete healing of scabs. Before the second and third treatment, 2D and 3D photographs will be taken. After each treatment, subjects will be asked to fill in the Therapy Comfort Questionnaire for the assessement of subjects' comfort during the treatments. After the last treament, subjects will receive Subject Satisfaction Questionnaire to record subjects' satisfaction with the treatment results.

At both follow-up visits, subjects will receive Subject Satisfaction Questionnaire to fill in, and 2D and 3D photographs will be taken.

Safety measures will include documentation of adverse events (AE) during and after the treatment procedures and at the follow-up visits, and if needed medical assistance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 30 years of age seeking treatment for improvement in skin quality and texture on face and neck
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Subjects willing and able to abstain from partaking in any facial or neck treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face and neck without makeup taken

Exclusion Criteria:

* Local bacterial or viral infection in the area to be treated
* Local acute inflammation in the area to be treated
* Impaired immune system caused by any immunosuppressive illness, disease or medication
* Isotretinoin and tretinoin-containing medication use in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants near the treatment area or neutral electrode
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis, and thrombosis)1
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Tuberculosis
* Hepatitis
* Febrile conditions
* Unwillingness/inability to not change their usual cosmetics and especially not to use anti-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* History of skin disorders, keloids, abnormal wound healing and dry or fragile skin
* Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks
* Neurotoxin/collagen/fat injections or other injected bio-material in the treated area within three months prior to the treatment
* Use of non-steroidal anti-inflammatory drugs one week before and after each treatment session
* Treating over tattoo or permanent make-up
* Treating over eyelids or the lips
* Patients with allergy to anesthetics
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Skin Quality Improvement Assessment | 12 months
  The primary efficacy outcome measure is aesthetic improvement 3 months post-treatment, assessed using 2D photographs on the Global Aesthetic Improvement Scale (GAIS), as well as the degree of clinical improvement determined by automated analysis of 3D photographs using the 3D analysis device's software. Improvement is considered an increase in the GAIS score, as well as in the score determined by the 3D analysis device's software.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 12 months
  To evaluate the safety of the BTL-785F device with the BTL-785-4-4 tip on the BTL-785-4 applicator for the improvement of skin quality and texture through monitoring of adverse reactions.
Satisfaction Assessed by the Subject Satisfaction Questionnaire | 12 months
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for the evaluation of satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last treatment, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' skin quality and overall facial appearance will vary from "strongly agree" to "strongly disagree".
Comfort Assessed by Therapy Comfort Questionnaire | 12 months
  The 5-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be given to subjects after each treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AboutSkin Dermatology & DermSurgery, Greenwood Village, Colorado
  - Capital Laser & Skin Care, Chevy Chase, Maryland
  - Boyd Beauty, Birmingham, Michigan